CLINICAL TRIAL: NCT04375072
Title: Combination Therapy of Home-based Transcranial Direct Current Stimulation and Mindfulness-based Meditation for Self-management of Clinical Pain and Symptoms in Older Adults With Knee Osteoarthritis
Brief Title: Home-based tDCS and Mindfulness-based Meditation for Self-management of Clinical Pain and Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hyochol Ahn, Dean & Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00003164; R01NR019051 (NIH); R01NR019051-03S1 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Osteo Arthritis Knee
Keywords: meditation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- active tDCS paired with active MBM, (Experimental)
  Interventions: Device: active tDCS paired with active MBM
- sham tDCS paired with active MBM (Active Comparator)
  Interventions: Device: sham tDCS paired with active MBM
- active tDCS paired with sham MBM (Active Comparator)
  Interventions: Device: active tDCS paired with sham MBM
- sham tDCS paired with sham MBM (Sham Comparator)
  Interventions: Device: sham tDCS paired with sham MBM

INTERVENTIONS:
Device: active tDCS paired with active MBM — Active tDCS with a constant current intensity of 2 milli ampere (mA) will be applied for 20 minutes per session daily for 2 weeks via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session daily for 2 weeks by a recorded meditation.
  Arms: active tDCS paired with active MBM,
Device: sham tDCS paired with active MBM — For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds during each 20-minute session, conducted daily for 2 weeks. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session daily for 2 weeks by a recorded meditation.
  Arms: sham tDCS paired with active MBM
Device: active tDCS paired with sham MBM — Active tDCS with a constant current intensity of 2 milli ampere (mA) will be applied for 20 minutes per session daily for 2 weeks via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. The sham MBM intervention will be delivered via a CD player that will look identical in both active and sham MBM.
  Arms: active tDCS paired with sham MBM
Device: sham tDCS paired with sham MBM — For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds during each 20-minute session, conducted daily for 2 weeks. The sham MBM intervention will be delivered via a CD player that will look identical in both active and sham MBM.
  Arms: sham tDCS paired with sham MBM

SUMMARY:
This clinical trial aims to evaluate whether a 2 week regimen of transcranial direct current stimulation (tDCS) paired with mindfulness-based meditation (MBM) can improve pain modulation, reduce clinical pain, and alleviate osteoarthritis (OA)-related symptoms in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* have symptomatic knee OA based on American College of Rheumatology clinical criteria
* have had knee OA pain in the past 3 months with an average of at least 30 on a 0-100 NRS for pain,
* can speak and read English
* have no plan to change medication regimens for pain throughout the trial

Exclusion Criteria:

* history of brain surgery, brain tumor, seizure, stroke, or intracranial metal implantation
* systemic rheumatic disorders, including rheumatoid arthritis,systemic lupus erythematosus, and fibromyalgia
* alcohol/substance abuse
* diminished cognitive function that would interfere with understanding study procedures (i.e., Mini-Mental Status Exam score ≤ 23)
* pregnancy or lactation
* prosthetic knee replacement or non-arthroscopic surgery to the affected knee
* hospitalization within the preceding year for psychiatric illness
* no access to a device that can be used for secure videoconferencing for real-time remote supervision.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyochol Ahn, PhD,RN,MSN, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 208 participants consented to participate in the study. However, 8 participants withdrew due to being unable to attend the remaining sessions and assessments.
Groups:
- active tDCS paired with active MBM: A 2mA current and mindfulness-based meditation are applied for 20 minutes
- sham tDCS paired with active MBM: A 2mA current is applied for 30 seconds, and mindfulness-based meditation is conducted for 20 minutes.
- active tDCS paired with sham MBM: A 2mA current is applied for 20 minutes, and mindfulness-based meditation without the specific instructions is conducted for 20 minutes.
- sham tDCS paired with sham MBM: A 2mA current is applied for 30 seconds, and mindfulness-based meditation without the specific instructions is conducted for 20 minutes.
Period: Overall Study
Arm/Group | active tDCS paired with active MBM | sham tDCS paired with active MBM | active tDCS paired with sham MBM | sham tDCS paired with sham MBM
Started | 53 | 53 | 50 | 52
Completed | 50 | 50 | 50 | 50
Not Completed | 3 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active tDCS Paired With Active MBM,: A transcranial direct current stimulation (tDCS) of 2mA is applied for 20 minutes, where a constant current of 2mA is delivered to the scalp through electrodes to modulate neural activity. Alongside this, mindfulness-based meditation is conducted for 20 minutes, focusing on cultivating awareness and concentration through practices such as breath observation and mindful awareness of thoughts and sensations. Both interventions are applied simultaneously, aiming to investigate their combined effects on brain function and mental state.
- Sham tDCS Paired With Active MBM: A 2mA transcranial direct current stimulation (tDCS) is applied for 30 seconds. Simultaneously, mindfulness-based meditation is conducted for 20 minutes, involving practices aimed at enhancing awareness and focus, such as observing the breath and maintaining attention to present-moment experiences.
- Active tDCS Paired With Sham MBM: A 2mA transcranial direct current stimulation (tDCS) is applied for 20 minutes, with a constant current of 2mA delivered through electrodes placed on the scalp to modulate neural activity in targeted brain regions. Simultaneously, mindfulness-based meditation without specific instructions is conducted for 20 minutes. In this meditation practice, participants are encouraged to focus on their breath and cultivate general awareness of their thoughts and sensations, without any particular guidance on how to direct their attention.
- Sham tDCS Paired With Sham MBM: A 2mA transcranial direct current stimulation (tDCS) is applied for 30 seconds. Simultaneously, mindfulness-based meditation without specific instructions is conducted for 20 minutes. In this practice, participants are encouraged to cultivate awareness and attention to their thoughts, feelings, and bodily sensations without any particular guidance or structured focus, allowing for an open-ended, self-directed meditation experience.
- Total: Total of all reporting groups
Arm/Group | Active tDCS Paired With Active MBM, | Sham tDCS Paired With Active MBM | Active tDCS Paired With Sham MBM | Sham tDCS Paired With Sham MBM | Total
Number analyzed (Participants) | 53 | 53 | 50 | 52 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.49 (7.74) | 67.19 (7.89) | 68.06 (7.42) | 68.88 (6.92) | 67.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 34 | 34 | 142
  Male | 19 | 13 | 16 | 18 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 2 | 11
  Not Hispanic or Latino | 51 | 50 | 46 | 50 | 197
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 3 | 6 | 20
  White | 44 | 41 | 43 | 43 | 171
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 4 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Rating Score (NRS) of Pain
Description: The Numeric Rating Scale (NRS) is a subjective measure of pain intensity. The NRS total score ranges from 0 (no pain) to 100 (most intense pain imaginable). Change in NRS = Week 2 (post-intervention) NRS - Baseline (pre-intervention) NRS. A decrease in NRS score indicates improvement.
Time Frame: baseline, week 2 (after 10 tDCS sessions)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | active tDCS paired with active MBM | sham tDCS paired with active MBM | active tDCS paired with sham MBM | sham tDCS paired with sham MBM
Number analyzed (Participants) | 53 | 53 | 50 | 52
units on a scale | -19.41 (19.76) | -7.16 (22.24) | -16.78 (17.90) | -6.20 (17.99)

2. Secondary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
Description: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): 26 question index to assess knee OA pain (0-20 scale), function (0-68 scale), and stiffness (0-8 scale). The total WOAMC score is the sum of the 3 sub scales for a total score range from 0-96. Change in total WOMAC score = Week 2 total WOMAC score - Baseline (pre-intervention) total WOMAC score. The lower change scores represents improvement in pain, movement, and stiffness.
Time Frame: baseline, week 2 (after 10 tDCS sessions)
Population: Comparison of WOMAC score changes between four groups at 2 weeks from baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- sham tDCS paired with active MBM: sham tDCS paired with active MBM: For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session daily for 2 weeks by a recorded meditation.
- active tDCS paired with sham MBM: active tDCS paired with sham MBM: Active tDCS with a constant current intensity of 2 mA will be applied for 20 minutes per session daily for 2 weeks via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. The sham MBM intervention will be delivered via a CD player that will look identical in both active and sham MBM.
- sham tDCS paired with sham MBM: sham tDCS paired with sham MBM: For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2 mA current for 30 seconds. The sham MBM intervention will be delivered via a CD player that will look identical in both active and sham MBM.
Arm/Group | active tDCS paired with active MBM, | sham tDCS paired with active MBM | active tDCS paired with sham MBM | sham tDCS paired with sham MBM
Number analyzed (Participants) | 53 | 53 | 50 | 52
units on a scale | -6.98 (13.27) | -7.90 (14.20) | -8.08 (13.39) | -4.50 (11.33)

ADVERSE EVENTS:
Time Frame: about 4 months
Groups:
- active tDCS paired with active MBM,: active tDCS paired with active MBM: Active tDCS with a constant current intensity of 2 milli ampere( mA)will be applied for 20 minutes per session daily for 2 weeks via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session daily for 2 weeks by a recorded meditation.
- sham tDCS paired with active MBM: sham tDCS paired with active MBM: For sham stimulation, the electrodes will be placed in the same positions as for active stimulation, but the stimulator will only deliver 2(milli ampere) mA current for 30 seconds. The meditation intervention will be applied simultaneously with tDCS for 20 minutes per session daily for 2 weeks by a recorded meditation.
Arm/Group | active tDCS paired with active MBM, | sham tDCS paired with active MBM | active tDCS paired with sham MBM | sham tDCS paired with sham MBM
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53 | 0/50 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/72/NCT04375072/Prot_SAP_001.pdf